CLINICAL TRIAL: NCT05346861
Title: Pyrotinib Rechallenge in Her2-positive Metastatic Breast Cancer Pretreated With Pyrotinib and Trastuzumab
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jian Zhang,MD, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YBCSG-21-01
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: HER2-positive Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Drug Therapy; pyrotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trastuzumab plus chemotherapy (Active Comparator)
  Interventions: Drug: Trastuzumab plus chemotherapy
- Pyrotinib in combination with Trastuzumab plus chemotherapy (Experimental)
  Interventions: Drug: Trastuzumab in combination with pyrotinib plus chemotherapy

INTERVENTIONS:
Drug: Trastuzumab plus chemotherapy — Trastuzumab: 8 mg/kg loading dose followed by 6 mg/kg, Q3W Chemotherapy regimen is chosen from the following: Vinorelbine, Gemcitabine, taxanes or Eribulin monotherapy Experimental: Pyrotinib +Trastuzumab + chemotherapy
  Arms: Trastuzumab plus chemotherapy
Drug: Trastuzumab in combination with pyrotinib plus chemotherapy — Pyrotinib: 400 mg po QD, Q3W Chemotherapy regimen is chosen from the following: Vinorelbine, Gemcitabine, taxanes or Eribulin monotherapy
  Arms: Pyrotinib in combination with Trastuzumab plus chemotherapy

SUMMARY:
Pyrotinib is an oral tyrosine kinase inhibitor targeting both HER-1 and HER-2 receptors. This study is a randomized, open-label, multi-center, parallel design study of the combination of pyrotinib, trastuzumab and chemotherapy versus trastuzumab and chemotherapy in HER2+ MBC patients, who have prior received trastuzumab and pyrotinib. Patients will be randomized in a 2:1 ratio to one of the following treatment arms. Arm A: pyrotinib + trastuzumab + chemotherapy, Arm B: trastuzumab + chemotherapy. Patients will receive either arm of therapy until disease progression, unacceptable toxicity, or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 and ≤75 years;
2. Pathologically confirmed HER2 positive patients with recurrence/ metastatic breast cancer: HER2 IHC 3+, or HER2 IHC 2+ and FISH detection gene amplification;
3. History of trastuzumab-containing chemotherapy in neoadjuvant, adjuvant or recurrence/ metastatic setting;
4. History of pyrotinib-containing chemotherapy in neoadjuvant or recurrence/ metastatic setting;
5. Previously reveived ≤2 systemic treatment in recurrence/ metastasis setting; (anti-HER2 ADCs such as T-DM1 is included in chemotherapy regimens, endocrine therapy alone is not included);
6. ECOG performance status of 0 to 1;
7. According to RECIST 1.1, at least one extracranial measurable lesion exists；
8. Signed informed consent.

Exclusion Criteria:

1. Patients with leptomeningeal metastasis or unstable brain metastasis;
2. History of neurological or psychiatric disorders;
3. Second malignancies within 5 years, except for cured skin basal cell carcinoma, carcinoma in-situ of uterine cervix and squamous-cell carcinoma;
4. Undergone major surgical procedures or significant trauma within 4 weeks prior to randomization, or expected to undergo major surgery.
5. Factors influencing the usage of oral administration (e.g. unable to swallow, chronic diarrhea and intestinal obstruction, etc.);
6. History of allergies to the drug components of this regimen;
7. History of Immunodeficiency, acquired or congenital immunodeficiency (HIV positive), history of organ transplantation;
8. Any other situations judged by investigator as not suitable for participating in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | approximately 8 months

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | approximately 8 months
Adverse Events (AEs) | From the first drug administration to within 28 days for the last treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Dai L, Gao T, Guo R, Chen Y, Wang J, Zhou S, Tang Y, Chen D, Huang S. Efficacy and safety of pyrotinib-based regimens in HER2 positive metastatic breast cancer: A retrospective real-world data study. Neoplasia. 2024 Oct;56:101029. doi: 10.1016/j.neo.2024.101029. Epub 2024 Jul 17. PMID 39024777